Numerical data was expressed as mean  $\pm$  standard deviation (SD) and qualitative data was expressed in percentage. The quantitative parameters was compared using student t test and the qualitative variables was compared using the Chi-square test. P value less than 0.05 was considered significant. Analyzed data was presented in the form of dummy tables, graphs, and charts. Data management, statistical analysis and data storage was done using Statistical Package for the Social Sciences (SPSS 21).